CLINICAL TRIAL: NCT02020096
Title: A Randomized Comparison of Ultrasound Plus Nerve Stimulator Guided Lumbar Plexus Block to Conventional Nerve Stimulator Guided Technique Using Winnie Approach
Brief Title: Ultrasound Plus Nerve Stimulator Versus Nerve Stimulator Guided Lumbar Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Wei Mei, Associate Professor, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TJMZK20131001
Record Dates: First submitted 2013-11-28; First posted 2013-12-24 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Knee Arthroscopy Surgery
Keywords: Lumbar plexus block; Ultrasound guidance; Nerve stimulator
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- U+N group (Experimental): Ultrasound and nerve stimulator guided lumbar plexus block combined with nerve stimulator guided sciatic block
  Interventions: Procedure: Ultrasound and nerve stimulator guided lumbar plexus block
- N group (Active Comparator): Nerve stimulator guided lumbar plexus block combined with nerve stimulator guided sciatic nerve block
  Interventions: Procedure: Nerve stimulator guided lumbar plexus block

INTERVENTIONS:
Procedure: Ultrasound and nerve stimulator guided lumbar plexus block — An insulated nerve block needle connected to a nerve stimulator that was delivering a current of 1.5 mA at a frequency of 2 Hz was then inserted in the long axis (in- plane) of the ultrasound transducer towards the the hypoechoic psoas compartment. If the quadriceps contraction which produces patella twitching was elicited with an initial current of 1.5mA,then the current should be reduced until contraction is still present between 0.3 to 0.5 mA .Afterward, the lumbar plexus nerve block was performed by using 30mL of 0.5% ropivacaine. Contraction should stop below a current of 0.3mA, otherwise intraneural needle position should be suspected.
  Arms: U+N group
Procedure: Nerve stimulator guided lumbar plexus block — The block was conducted following traditional Winnie approach. The accepted end point for the lumbar plexus is stimulation of the femoral nerve component, observed by contraction of the quadriceps muscle. Quadriceps contraction which produces patella twitching should be sought with an initial current of 1.5mA, and once elicited the current should be reduced until contraction is still present between 0.3 to 0.5 mA. Afterward, the lumbar plexus nerve block was performed by using 30mL of 0.5% ropivacaine. Contraction should stop below a current of 0.3mA, otherwise intraneural needle position should be suspected.
  Arms: N group

SUMMARY:
Ultrasound imaging, an effective tool to localize peripheral nerves, may facilitate block performance. It allows direct visualization of nerve structures, needle guidance in real-time to the target, and observation of local anesthetic diffusion. Some case series have demonstrated significantly faster onset time for interscalene blocks, supraclavicular blocks and axillary brachial plexus blocks under ultrasound than with conventional techniques. Ultrasound guidance also enhances the quality of popliteal sciatic nerve block at the popliteal fossa compared with single injection, nerve stimulator-guided block using either a tibial or peroneal endpoint. Despite this impressive profile, the application of the ultrasound for lumbar plexus blocks has not been studied extensively. It is likely that lumbar plexus block (LPB) combined with either a sciatic nerve block or sedation or both is equivalent to general anesthesia and neuraxial anesthesia for knee arthroscopy. The lumbar plexus block is traditionally performed using surface anatomical landmarks and nerve stimulation. Ultrasound imaging of the anatomy relevant for LPB is challenging because of its deep anatomic location and the "acoustic shadow" of the overlying transverse processes. Recently, Karmakar M.K. etc. has demonstrated that a paramedian transverse scan (PMTS) of the lumbar paravertebral region with the ultrasound beam being insonated through the intertransverse space (ITS) and directed medially toward the intervertebral foramen (PMTS-ITS) may overcome the problem of the "acoustic shadow" and allow clear visualization of the anatomy relevant for LPB. However, the application of a PMTS-ITS used for lumbar plexus blocks has not been studied extensively and its advantages are not validated in a clinical study. Thus, we designed this prospective, randomized, subject and assessor blinded, parallel-group, active-controlled study to compare a PMTS ultrasound-guided lumbar plexus block combined with nerve stimulation and a conventional technique on time required to readiness for surgery in patients undergo knee arthroscopy surgery.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Age 18-70yr
* American Society of Anesthesiologists physical status I-II
* Patients scheduled to undergo knee arthroscopy surgery
* Ultrasound visibility score equal or great than 10

Exclusion Criteria:

* Body mass index more than 35 kg/m²
* Pregnant or lactating women
* Allergy to local anesthetics
* Coagulopathy, on anticoagulants
* Malignancy or infection at puncture site
* Significant peripheral neuropathy or diabetic peripheral neuropathy
* Language barrier
* Neuropsychiatric disorder
* Severe cardiac or respiratory diseases
* Pathology or previous surgery or trauma to the lower limb
* Analgesics intake, history of substance abuse
* History of spinal surgery or deformity
* Ultrasound visibility score less than 10
* Participating in the investigation of another experimental agent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Onset time of sensory block to cold and pinprick | up to 40 min after ropivacaine injection
  Onset time of sensory block (cold/pinprick), defined as time interval from completion of local anesthetic injection to the achievement of complete sensory block (defined as no sensation in three major branches including the femoral nerve, the lateral femoral cutaneous nerve and the obturator nerve) .

SECONDARY OUTCOMES:
Total ultrasound visibility score (UVS) | 30 min before and 5 min after lumbar plexus block
  The independent observer attempted to visualize 10 paravertebral structures in images of the ultrasound scans from the patients
Performance time of block | up to 20 min after needle insertion
  Performance time of block is the preparing time and procedure time. Preparing time (defined as the time from the beginning of the sterile preparation right before the first needle contact with the skin). Procedure time (time between the insertion of the needle and the end of local anesthetic injection)
Number of needle passes during block | up to 20min after needle insertion
  Number of needle passes during block
Minimal stimulating current of the needle | up to 20min after needle insertion
  All peripheral nerve blocks were performed by the same anesthesiologist with an 100-mm insulated stimulating needle attached to a nerve stimulator. The intensity of the stimulating current, initially set to deliver 1 to 1.5 mA (0.1ms, 2Hz), was gradually decreased to <0.5 mA while the appropriate motor response was maintained.
  For sciatic block, the targeted evoked motor response was plantar flexion of the foot. For lumbar plexus block, quadriceps muscle motor response was targeted.Contraction should stop below a current of 0.2mA, otherwise intraneural needle position should be suspected and the needle should be withdraw and readjusted. The Minimal stimulating current ( intensity of the current when the needle was considered to be adequately positioned) finally demonstrated on nerve stimulator was recorded, then ropivacaine was injected slowly after careful intermittent aspirations.
Onset time of motor block | up to 40min after ropivacaine injection
  onset time of motor block, defined as time interval from completion of local anesthetic injection to the achievement of satisfied motor block (defined as a Modified Bromage scale equal to 3).
Incidence of paresthesia during block | up to 20min after needle insertion
  Incidence of paresthesia during block reported by patients
Incidence of accidental vascular puncture | up to 20min after needle insertion
  Incidence of accidental vascular puncture, defined as blood by aspiration.
Changes of muscle strength of quadriceps femoris and adductors | up to 40min after ropivacaine injection
  Muscle strength of quadriceps femoris and adductors was measured with hand-held dynamometer (HHD, Hogan Health Industries, MicroFET3) during knee extension and hip adduction.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Mei, MD., PhD., Principal Investigator — Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology; Yuke Tian, MD., PhD., Study Chair — Department of Anesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China